CLINICAL TRIAL: NCT04621617
Title: Midodrine and Albumin in Patients With Refractory Ascites. A Randomised Controlled Trial.
Brief Title: Midodrine and Albumin in Patients With Refractory Ascites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor and Head, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC-06/2020-1691
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Refractory Ascites
MeSH Terms: conditions — Ascites | interventions — Albumins; Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Albumin + Midodrine + SMT (Active Comparator): Human albumin plus oral midodrine
  Interventions: Drug: Albumin; Drug: Midodrine; Drug: Standard medical therapy (SMT)
- Albumin + SMT (Active Comparator): Human albumin plus placebo of midodrine
  Interventions: Drug: Albumin; Drug: Standard medical therapy (SMT)
- SMT (Placebo Comparator): standard medical therapy plus placebo of midodrine
  Interventions: Drug: Standard medical therapy (SMT)

INTERVENTIONS:
Drug: Albumin — Human albumin will be administered by intravenous infusion at a dose of 1.5 gm/kg/week for 2 weeks followed by HA 40 grams every 7days
  Arms: Albumin + Midodrine + SMT; Albumin + SMT
Drug: Midodrine — Oral Midodrine will be given at a dose of 7.5 mg three times in a day
  Arms: Albumin + Midodrine + SMT
Drug: Standard medical therapy (SMT) — SMT will include nutritional support, rifaximin, lactulose or lactitol, diuretics, SBP prophylaxis with norfloxacin, restriction of sodium, multivitamins, and other supportive measures as deemed necessary. LVP will be done as needed. Patients on non-selective beta blockers will continue to do so with dose modifications/withdrawal as per Baveno VI guidelines.

SUMMARY:
Refractory ascites is seen in 5-10% of patients with cirrhosis.Decompensated cirrhosis with refractory ascites has a mortality rate of around 40% in a year and a median survival of 6 months.Portal hypertension and splanchnic vasodilation are major factors in the development of ascites.The treatment of refractory ascites involves salt restriction, diuretics, large volume paracentesis (LVP), transjugular Intrahepatic Portosystemic shunt (TIPS) and Liver Transplantation (LT). Currently the only curative treatment is LT. However, LT is limited due to organ shortage and high cost.

Long-term human albumin (HA) administration in patients with uncomplicated and refractory ascites, has shown to improve survival or delay the complications of cirrhosis. Midodrine, an oral α1- adrenergic agonist has been used in refractory ascites with variable results. However, there is no study on the use of long term Midodrine and HA in patients with refractory ascites. Therefore, we plan to study the effect of long term midodrine and HA in patients with refractory ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years
2. Refractory ascites in cirrhosis of any etiology

Exclusion Criteria:

1. Mixed ascites: cirrhosis plus another cause of ascites
2. Gastrointestinal bleed within 7 days of enrolment.
3. Presence of hepatorenal syndrome
4. Hepatic encephalopathy grade 2 or higher
5. Infection within 1 month preceding the study
6. Cardiovascular disease (ejection fraction < 35% or abnormal ECG) or arterial hypertension (BP > 140/90 mm of Hg)
7. Abnormal urine analysis with proteinuria > 500 mg/24 hour or 50 red blood cells/high power field, or granular casts or ultrasonographic evidence of intrinsic renal disease
8. Presence of hepatocellular carcinoma or portal vein thrombosis
9. Treatment with drug with known effects on systemic and renal hemodynamics within 7 days of inclusion excepting beta-blockers
10. Patient not willing for study.
11. Patient opting for liver transplantation/ transjugular intrahepatic portosystemic shunt

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with control of ascites at 1 year | 1 year
  Control of ascites will be defined as-
  * Complete response will be total absence of ascites.
  * Partial response as presence of ascites not requiring paracentesis
  * Non response will be defined as persistence of severe ascites requiring paracentesis.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) measured by modified diet in renal disease 6 (MDRD6) formula at 3 months intervals | 1 year
  eGFR will be measured using MDRD6 formula
Changes in concentration of albumin at 3 months intervals | 1 year
  Change in concentration of serum albumin (g/dl)
Change in model for end stage liver disease (MELD) score | 1 year
  Change in MELD score. The MELD score incorporates the variables of serum bilirubin, creatinine and Internation Normalised Ratio (INR). Higher MELD score indicates worse prognosis
Change in mean arterial pressure at 3 months interval | 1 year
  Change in mean arterial pressure (mm of Hg) will be noted
Changes in serum and 24- hour urine sodium | 1 year
  Serum and urine sodium concentration will be measured in meq/L
Incidence of spontaneous bacterial peritonitis (SBP) and other infections | 1 year
  The diagnosis of SBP will be based on neutrophil count in ascitic ﬂuid of >250/mm3 as determined by microscopy and positive ascitic fluid culture or >250 /mm3 with negative culture called as culture negative neutrocytic ascites.20 Other infections will be diagnosed as per CDC criteria.
Number of patients who develop paracentesis induced circulatory dysfunction (PICD) | 1 year
  PICD will be defined as an increase in plasma renin activity (PRA) of >50% of the pre-treatment value to a level > 4ng/ml/hr on 6th day after paracentesis
Number of patients who develop hyponatremia | 1 year
  Hyponatremia will be defined using serum sodium concentrations of <130meq/L.
Change in Child-Turcotte-Pugh (CTP) score | 1 year
  Change in CTP score. The CTP score incorporates the variables of serum bilirubin, albumin, prothrombin time-INR, grade of ascites and hepatic encephalopathy. The score ranges from 5-15 and a higher score portends a worse prognosis
Number of patients who develop hypokalemia | 1 year
  Hypokalemia will be defined using serum potassium levels <3 meq/L
Number of patients who develop hyperkalemia | 1 year
  hyperkalemia will be defined using serum potassium levels >6 meq/L

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, MD, DM, Principal Investigator — PGIMER, Chandigarh

IPD SHARING:
Plan to Share IPD: No